CLINICAL TRIAL: NCT03639766
Title: The Effect of Abobotulinum Toxin A on the Symptoms of Raynaud's Phenomenon, a Double-Blind Randomized Placebo-Controlled Trial
Brief Title: The Effect of Abobotulinum Toxin A on the Symptoms of Raynaud's Phenomenon
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Time and resource constraints
Sponsor: University of Central Florida (Other)
Responsible Party: Principal Investigator, David Weinstein, Assistant Professor of Dermatology, University of Central Florida
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BIO-18-14092
Record Dates: First submitted 2018-08-17; First posted 2018-08-21 (Actual); Results first posted 2021-06-30 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Raynaud Phenomenon
Keywords: Raynaud Phenomenon; AbobotulinumtoxinA
MeSH Terms: conditions — Raynaud Disease | interventions — abobotulinumtoxinA; Saline Solution

STUDY DESIGN:
Intervention Model Description: This is a two-arm parallel assignment involves two groups of participants. One group/hand receives the abobotulinum toxin A, and the other group/hand receives a saline solution (control).
Who Masked: Participant, Investigator
Masking Description: This is a double-blind placebo-controlled trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Abobotulinum toxin A (Experimental): Injection of 300 units of abobotulinum toxin A in 10 ml of non-bacteriostatic normal saline to chosen hand.
  Interventions: Drug: AbobotulinumtoxinA
- Saline solution (Placebo Comparator): Injection of 10 ml of non-bacteriostatic normal saline to chosen hand.
  Interventions: Other: Saline solution

INTERVENTIONS:
Drug: AbobotulinumtoxinA — AbobotulinumtoxinA reconstituted in non-bacteriostatic saline solution
  Arms: Abobotulinum toxin A
Other: Saline solution — Non-bacteriostatic saline solution
  Arms: Saline solution

SUMMARY:
This study aims to investigate the effect of abobotulinum toxin A on the symptoms of Raynaud's phenomenon.

DETAILED DESCRIPTION:
This prospective double-blind randomized control trial seeks to compare a single formulation of BoNT, aboboutlinum toxin A (Dysport), to a placebo saline group, studying the effect of BoNT on Raynaud's symptoms among a more diverse population to provide insight into the patients most likely to benefit from BoNT.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adult between 18 and 80 years of age
* Must have health insurance
* Must have a current diagnosis of Raynaud's phenomenon

Exclusion Criteria:

* Allergy to abobotulinum toxin A or its components
* Diagnosis of myasthenia gravis
* Previously received abobotulinum toxin vaccine
* Previously undergone upper extremity vascular surgery (including surgical sympathectomy)
* Currently receiving aminoglycoside antibiotics
* Received abobotulinum toxin A treatment in either hand in the past 6 months
* Pregnant women
* Women currently breastfeeding
* Current tobacco smoker (use in the past 12 months)
* Unable to read and speak English
* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-08-31 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UCF Health Lake Nona Office, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study had to be close early due to lack of support and time resulting in a lower number of participants than hoped for.
Groups:
- All Study Participants: All study participants received an injection of Abobotulinum Toxin A into one hand. They received an injection of saline in the other hand.
  The Abobotulinum Toxin A injection solution consisted of 300 units in 10 ml of non-bacteriostatic normal saline.
  The saline injection consisted of 10 ml of non-bacteriostatic normal saline.
Period: Overall Study
Arm/Group | All Study Participants
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Study Participants
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Raynaud's Condition Score
Description: Raynaud's Condition Score is a validated outcome measure used to assess a person's functionality owing to their Raynaud's symptoms. 0 to 10, with 0 being no symptoms and 10 being more severe symptoms of Raynaud's.
Time Frame: 12 months
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Abobotulinum Toxin A | Saline Solution
Number analyzed (Participants) | 3 | 3
score on a scale
  Baseline | 1.3 [0 to 4] | 1.3 [0 to 4]
  3 Months | 3 [1 to 4] | 0.67 [0 to 2]
  9 Months | 1 [0 to 3] | 1 [0 to 3]
  12 Months | 1.4 [0 to 3.3] | 0.6 [0 to 1]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Abobotulinum Toxin A | Saline Solution
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 2/3 | 0/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abobotulinum Toxin A (N=3) | Saline Solution (N=3)
Hand Weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) — Hand muscle weakness

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-09-26): https://cdn.clinicaltrials.gov/large-docs/66/NCT03639766/Prot_SAP_000.pdf
  • Informed Consent Form (2019-05-21): https://cdn.clinicaltrials.gov/large-docs/66/NCT03639766/ICF_001.pdf